CLINICAL TRIAL: NCT02570698
Title: Collection and Characterization of Premature Infants Feces for Identification of Factors Contributing to Skin Irritation
Brief Title: BM Collection From NICU Infants for Composition
Status: Completed | Type: Observational
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 500-15-0001
Record Dates: First submitted 2015-09-30; First posted 2015-10-07 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Diaper Dermatitis
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to collect feces from premature infants over a five weeks period to characterize its composition. Metabolomics, Proteomics, Genomics and Microbiome analyses and cell-based assays will be performed to identify individual components present in feces, which may contribute to the onset of irritation in the diapered area of premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Infant's parent(s)/legal guardian(s) must be fluent in English or Spanish, willing and able to read, understand, and sign the informed consent form (ICF).
* Infants (male or female) who are equal or less than a gestational age of 30 weeks + 4 days.

Exclusion Criteria:

* Any medical condition which, in the opinion of the principal investigator, may compromise infant's safety.
* Any underlying chronic skin conditions. However, infants may participate in the study with a rash in the diapered area if, in the opinion of the principal investigator, this does not compromise infant's safety.

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who are equal or less than a gestational age of 30 weeks + 4 days
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12-07 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Composition of proteins (ug/uL) in premature infant feces | 0 to 5 weeks
  This is an observational study where fecal samples will be collected twice each week for 5 weeks from enrolled patients. Primary analysis will consist of identification and quantification proteins present in samples.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Eichenfield, MD, Principal Investigator — UCSD Rady Children's Hospital
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

REFERENCES:
- [Background] Stamatas GN, Nikolovski J, Mack MC, Kollias N. Infant skin physiology and development during the first years of life: a review of recent findings based on in vivo studies. Int J Cosmet Sci. 2011 Feb;33(1):17-24. doi: 10.1111/j.1468-2494.2010.00611.x. Epub 2010 Aug 30. PMID 20807257
- [Background] Kalia YN, Nonato LB, Lund CH, Guy RH. Development of skin barrier function in premature infants. J Invest Dermatol. 1998 Aug;111(2):320-6. doi: 10.1046/j.1523-1747.1998.00289.x. PMID 9699737
- [Background] Andersen PH, Bucher AP, Saeed I, Lee PC, Davis JA, Maibach HI. Faecal enzymes: in vivo human skin irritation. Contact Dermatitis. 1994 Mar;30(3):152-8. doi: 10.1111/j.1600-0536.1994.tb00696.x. PMID 8187514
- [Background] Buckingham KW, Berg RW. Etiologic factors in diaper dermatitis: the role of feces. Pediatr Dermatol. 1986 Feb;3(2):107-12. doi: 10.1111/j.1525-1470.1986.tb00499.x. PMID 3513143
- [Background] Visscher, Marty O. Recent advances in diaper dermatitis: etiology and treatment. Pediatric Health 3(1):81-98, 2009
- [Background] Visscher M, Narendran V. Neonatal Infant Skin: Development, Structure and Function. Newborn and Infant Nursing Review 14(4):135-141, 2014.
- [Background] Stamatas GN, Tierney NK. Diaper dermatitis: etiology, manifestations, prevention, and management. Pediatr Dermatol. 2014 Jan-Feb;31(1):1-7. doi: 10.1111/pde.12245. Epub 2013 Nov 14. PMID 24224482
- [Background] Bruderer R, Bernhardt OM, Gandhi T, Miladinovic SM, Cheng LY, Messner S, Ehrenberger T, Zanotelli V, Butscheid Y, Escher C, Vitek O, Rinner O, Reiter L. Extending the limits of quantitative proteome profiling with data-independent acquisition and application to acetaminophen-treated three-dimensional liver microtissues. Mol Cell Proteomics. 2015 May;14(5):1400-10. doi: 10.1074/mcp.M114.044305. Epub 2015 Feb 27. PMID 25724911